CLINICAL TRIAL: NCT06598137
Title: Multicenter, Prospective Study to Examine Pigmented, Non-pigmented, Tumorous and Inflammatory Lesions of the Skin With Regard to Cut Margin Control, Differentiation, Grading and Tumor Thickness Using Confocal Laser Microscopy
Brief Title: Study to Examine Lesions of the Skin Using Confocal Laser Microscopy
Status: Active, not recruiting | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Maximilian Deußing, Principal Investigator, LMU Klinikum
Other Study IDs: 23-0393
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Benign Skin Tumor; Basal Cell Carcinoma; Melanoma; Squamous Cell Cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Melanoma; Neoplasms, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ex vivo confocal laser microscopy — Using ex-vivo confocal laser scanning microscopy, a reliable statement can be made about the extent, histological structure and possible significance of a skin change without having to send tissue samples for demanding and lengthy histological examinations.

SUMMARY:
Using ex-vivo confocal laser scanning microscopy, a reliable statement can be made about the extent, histological structure and possible significance of a skin change without having to send tissue samples for demanding and lengthy histological examinations.

DETAILED DESCRIPTION:
Using ex-vivo confocal laser scanning microscopy, a reliable statement can be made about the extent, histological structure and possible significance of a skin change without having to send tissue samples for demanding and lengthy histological examinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign and malignant skin tumors

Exclusion Criteria:

* Patients unable to consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with benign and malignant skin tumors
Sampling Method: Probability Sample
Enrollment: 645 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Reaching the planned number of patients >640 | approx. 1-4 years
  Reaching the planned number of patients >640

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Dermatology and Allergy LMU Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No